CLINICAL TRIAL: NCT04071808
Title: Changes of Plasma Orphanin and Norepinephrine Levels in Patients With Painless Myocardial Ischemia and Diabetes Mellitus.
Brief Title: Painless Myocardial Ischemia in Diabetic Patients.
Status: Completed | Type: Observational
Sponsor: Second Hospital of Shanxi Medical University (Other)
Responsible Party: Principal Investigator, Zheng Guo, professor, Second Hospital of Shanxi Medical University
Other Study IDs: hanyi20190825
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Painless Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Coronary angiography group: In diabetic patients without symptoms of myocardial ischemia, coronary angiography showed no stenosis or stenosis less than 75%.
  Interventions: Diagnostic Test: ELISA Test
- Coronary angiographic stent implantation group: Coronary angiographic stenosis was more than 75% in diabetic patients without myocardial ischemia symptoms, and coronary stents were implanted.
  Interventions: Diagnostic Test: ELISA Test

INTERVENTIONS:
Diagnostic Test: ELISA Test — The levels of orphanin and norepinephrine in blood of diabetic patients with painless myocardial ischemia requiring interventional therapy and diabetic patients without interventional therapy were measured.

SUMMARY:
This study aims to investigate the relationship between the concentrations of blood orphanin, norepinephrine and the morbidity of painless myocardial ischemia in patients with diabetes mellitus. Hopefully, the biomarker(s) in the blood of diabetic patients can be found for screening high risk patients in the diabetes sufferers to prevent the painless myocardial ischemia.

ELIGIBILITY:
Inclusion Criteria:

* Subject has diabetes

Exclusion Criteria:

* History of myocardial ischemia
* Symptoms of myocardial ischemia（ECG changes except）

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Blood orphanin content | 24 hours
  Blood orphanin levels in painless diabetic patients with myocardial ischemia requiring interventional therapy and diabetic patients without interventional therapy.
Blood norepinephrine content | 24 hours
  Blood norepinephrine levels in diabetic patients with painless myocardial ischemia requiring interventional therapy and diabetic patients without interventional therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Second of Shanxi Medical University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication.